CLINICAL TRIAL: NCT05666648
Title: Comparison of Sitz Bath and no Sitz Bath Treatments in Patients With Acute Anal Fissure
Brief Title: Sitz Bath vs no Sitz Bath in Acute Anal Fissure Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Combined Military Hospital Quetta (Other)
Responsible Party: Principal Investigator, Dr Zeeshan Ayub, Associate Professor, Combined Military Hospital Quetta
Other Study IDs: IRB/851/CMH Quetta
Record Dates: First submitted 2022-12-11; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Pain, Postoperative
Keywords: Acute anal fissure, pain, sitz bath
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sixty patients completed trial in two groups
  Interventions: Other: Sitz Bath

INTERVENTIONS:
Other: Sitz Bath — Individual patients were randomized to either receive 'sitz baths' or 'no sitz baths' treatment for 4 weeks. Patients were asked to have 'sitz bath' once in morning and again at bedtime, after each week pain scores and healing of fissure were assessed. Main outcome measures were validated

SUMMARY:
To compare the efficacy of 'sitz bath' and 'no sitz bath' treatment in terms of pain improvement, rate of cure and fissure healing in Acute Anal Fissure.

DETAILED DESCRIPTION:
ABSTRACT Objective To compare the efficacy of 'sitz bath' and 'no sitz bath' treatment in terms of pain improvement, rate of cure and fissure healing in Acute Anal Fissure.

Study Design Randomized Controlled Trial Place and Duration of Study Department of Surgery Combined Military Hospital, Quetta, from15 January 2019 to 15 August 2021.

Patients and Methods Individual patients were randomized to either receive 'sitz baths' or 'no sitz baths' treatment for 4 weeks. Patients were asked to have 'sitz bath' once in morning and again at bedtime, after each week pain scores and healing of fissure were assessed. Main outcome measures were validated.

Keywords Acute anal fissure, pain, sitz bath

ELIGIBILITY:
Inclusion Criteria:

* Patients of acute anal fissure of both genders between 18 to 60 years

Exclusion Criteria:

* While the patients with history of recurrent fissure, chronic anal fissure, pregnant woman and patients who were operated previously for any anorectal pathology were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of acute anal fissure of both genders between 18 to 60 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
healing of fissure | four weeks
  healing of fissure after 4 weeks sitz bath

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Ayub, FCPS, Study Director — CMH Quetta
Locations (1):
- Khalid Pervaiz, Quetta, Pakistan

IPD SHARING:
Plan to Share IPD: No
Plan to work further